CLINICAL TRIAL: NCT02719249
Title: Fabry Disease Prevalence in End-stage Renal Disease (ESRD) Patients on Dialysis or Transplant in West of France
Brief Title: Fabry Disease Screening in ESRD Patients in West of France
Acronym: SNOUFY
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC14-9733
Record Dates: First submitted 2016-03-21; First posted 2016-03-25 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-02

CONDITIONS: ESRD
Keywords: ESRD; Fabry disease
MeSH Terms: conditions — Kidney Failure, Chronic; Fabry Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Men with ESRD on dialysis or transplant
  Interventions: Other: Dried blood spot test

INTERVENTIONS:
Other: Dried blood spot test

SUMMARY:
Screening of Fabry disease in end-stage renal disease (ESRD) patients on dialysis or transplant in west of France.

DETAILED DESCRIPTION:
Detection of Fabry disease is done by dried blood spot test, in dialyzed and transplanted men, who reached ESRD for vascular or unknown disease and were not previously screened.

ELIGIBILITY:
Inclusion Criteria:

* Men less than 70 years old
* ESRD treated by dialysis or kidney graft in one of the 4 following regions : Bretagne, Centre, Pays de la Loire and Poitou-Charentes
* For unknown nephropathy OR vascular nephropathy and/or diabetic nephropathy unproved by biopsy
* Agreeing freely to participate in the study

Exclusion Criteria:

* Men less than 18 years old
* Persons subject to major legal protection (safeguarding justice, guardianship, trusteeship), persons deprived of liberty.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: End-stage renal disease patients
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2016-01; Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
To detect Fabry disease by dried blood spot test, in dialyzed and transplanted men, who reached ESRD for vascular or unknown disease and were not previously screened | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No